CLINICAL TRIAL: NCT05098899
Title: Interventions Using Genomics-based Strategies (InGeSt) Towards Enhanced Nutrition Recommendations: A Proof-of-concept RCT for the DNA-based Nutrition and Lifestyle Recommendations in Overweight and Obese Filipino Adults
Brief Title: MyGeneMyDiet Trial for Weight Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Food and Nutrition Research Institute, Philippines (Other Government)
Responsible Party: Principal Investigator, Jacus Nacis, Senior Science Research Specialist, Food and Nutrition Research Institute, Philippines
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 19-003-00-00000-2-12-6-2021
Record Dates: First submitted 2021-10-20; First posted 2021-10-28 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2024-09

CONDITIONS: Overweight and Obesity
Keywords: Overweight; Obesity; Nutritional Genomics; Nutrigenomics; DNA-based nutrition advice; Genotype-based nutrition advice
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MyGeneMyDiet® Recommendations for Weight Management (Experimental): A set of nutrition and lifestyle advice for weight management derived from genetic information
  Interventions: Genetic: MyGeneMyDiet® Recommendations for Weight Management
- Usual Standard of Care for Weight Management (Active Comparator): A set of standard nutrition and lifestyle advice for weight management without genetic information
  Interventions: Other: Usual Standard of Care for Weight Management

INTERVENTIONS:
Genetic: MyGeneMyDiet® Recommendations for Weight Management — This group will receive Nutrition and Lifestyle recommendation based on SNPs known to have an impact to body weight and body composition, and responses to physical activity and dietary fat intake
  Arms: MyGeneMyDiet® Recommendations for Weight Management
Other: Usual Standard of Care for Weight Management — This group will receive the conventional and standard nutrition lifestyle recommendation for weight management
  Arms: Usual Standard of Care for Weight Management

SUMMARY:
The study aims to determine if genotype-based nutrition and lifestyle advice is effective for the management of overweight and obesity among Filipino adults compared to the usual standard of care.

DETAILED DESCRIPTION:
The primary objective of the study is to determine if providing a nutrition and lifestyle advice with genetic information can promote the attainment of 5-10% weight loss, and improvements on body mass index, waist circumference, and body fat percentage among Filipino adults with overweight and obesity. Additionally, changes in dietary intake, eating behaviour, physical activity level, biochemical parameters (HbA1c and blood lipid profile), motivation for weight loss, and knowledge and perceptions on nutrigenomics and genetic testing will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese Filipino adults who signify a willingness to participate in the study
* With BMI equal to 25.0 but not more than 40 kg/m2
* Apparently healthy (fasting blood glucose, lipid profile, and blood pressure within the normal range to pre-disease state)
* Normal thyroid hormone levels in the blood
* Normal blood cortisol level
* Carriers of at least one of the risk alleles of FTO rs9939609, UCP1 rs1800592, and TCF7L2 rs7903146

Exclusion Criteria:

* Elevated levels of fasting blood glucose, blood lipids, and blood pressure
* Elevated levels of thyroid hormones, and cortisol level
* Self-reported/history of heart disease
* Participation in a weight loss program or adherence to restrictive /therapeutic diet in the past 3 month
* Self-reported of recent weight changes greater or less than 3.0 kg
* Planned or recent bariatric surgery
* Consumption of weight-altering medications and/or nutritional supplements that promote weight gain/loss in the past 6 months
* Clinical diagnosis of any mental disorder and current use of any mental health medications
* Pregnant, nursing, or with self-declared intention to become pregnant
* Any health condition that may put the participant at risk
* Current and anticipated enrolment in another research study during the course of the trial

Ages: 19 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
5% weight loss | 24 weeks
  Attainment of 5% weight loss
10% weight loss | 48 weeks
  Attainment of 10% weight loss
Body mass index | 24 weeks
  Changes in BMI
Waist circumference | 24 weeks
  Changes in waist circumference
Body fat percentage | 24 weeks
  Changes in body fat percentage

SECONDARY OUTCOMES:
Dietary intake | 24 weeks
  Improvements in dietary intake
Eating behavior | 24 weeks
  Improvements in eating behavior
Physical activity level | 24 weeks
  Improvements in physical activity level
Glycated haemoglobin (HbA1c) | 24 weeks
  Changes in HbA1c
Blood lipid profile (TC, LDL-C, HDL-C, Triglycerides) | 24 weeks
  Changes in TC, LDL-C, HDL-C, Triglycerides
Motivation for weight loss | 24 weeks
  Stages and motivation for weight loss
Knowledge and perceptions | 24 weeks
  Knowledge and perceptions in nutrigenomics and genetic testing

CONTACTS AND LOCATIONS:
Overall Officials: Jacus S Nacis, MBAH, Principal Investigator — Department of Science and Technology-Food and Nutrition Research Institute (DOST-FNRI)
Locations (1):
- Department of Science and Technology-Food and Nutrition Research Institute, City of Taguig, National Capital Region, Philippines

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nacis JS, Labrador JPH, Ronquillo DGD, Rodriguez MP, Dablo AMFD, Frane RD, Madrid ML, Santos NLC, Carrillo JJV, Fernandez MG, Gonzales GBL. A study protocol for a pilot randomized controlled trial to evaluate the effectiveness of a gene-based nutrition and lifestyle recommendation for weight management among adults: the MyGeneMyDiet(R) study. Front Nutr. 2023 Aug 22;10:1238234. doi: 10.3389/fnut.2023.1238234. eCollection 2023. PMID 37674889